CLINICAL TRIAL: NCT05146557
Title: Associations Between Obesity, Dental Caries, Erosive Tooth Wear and Periodontal Disease in Adolescents: A Case Control-study
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 670201423056
Record Dates: First submitted 2019-12-09; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Obesity, Childhood; Tooth Wear; Tooth Erosion; Dental Caries; Dental Plaque; Gingivitis
Keywords: Tooth wear
MeSH Terms: conditions — Obesity; Pediatric Obesity; Tooth Wear; Tooth Erosion; Dental Caries; Dental Plaque; Gingivitis | interventions — Diagnosis, Oral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Obese adolescents: BMI above the 97th percentile + 2.17 to+2.18 SDS
  Interventions: Other: Dental examination
- Group Normal weight adolescents: BMI between the 10th and 90th percentile -1.64 to +1.64 SDS
  Interventions: Other: Dental examination

INTERVENTIONS:
Other: Dental examination — In this cross sectional observational study only Dental examination and a self response survey was applied.

SUMMARY:
Objectives To compare oral health (dental caries, periodontal status, and erosive tooth wear (ETW)), diet and oral hygiene habits between obese and normal weight adolescents, and to explore possible risk associations.

Materials and Methods In this case-control study, a convenient sample of 81 obese adolescents (age range 11-18) from a rehabilitation centre, and 81 age-sex-matched normal weight adolescents were selected. Groups were defined using the Body Mass Index and growth curves for Flemish. Oral health was measured using DMFT, gingival, plaque and BEWE index. A validated questionnaire was utilized to assess diet and oral hygiene habits.

DETAILED DESCRIPTION:
Participants and ethical aspects For this case-control study, a total of 162 adolescents residing in Belgium were examined between July 2015 and October 2015.

Height and weight were measured to calculate the Body Mass Index (BMI) of the participants. Obese and normal weight groups were defined using the BMI according to the European Childhood Obesity Group (ECOG) and the growth curves for Flemish boys and girls (2-20years). Only the participants with obesity were included in the case group (having a BMI above the 97th percentile + 2.17 to+2.18 SDS), whereas only the participants with normal weight were included in the control group (BMI between the 10th and 90th percentile -1.64 to +1.64 SDS).

Clinical examination Anthropometrical and dental examinations were performed in the educational institutions. Before scoring, dental surfaces were dried using sterile gauze. Standard illumination (LED head lamps), sterile number five mouth mirrors and CPI periodontal probes (WHO 1997) were used. Caries experience was screened using DMFT index (Decayed, Missing, Filled Teeth) with a subdivision for D1 (early caries, 'white spots'), D2 (enamel caries) or D3 (dentine caries). The periodontal status was evaluated by measuring the Gingivitis index (Silness and Loë, 1963), Plaque index (Silness and Loë, 1964) and the presence of periodontal pockets (≥4mm) in all Ramfjord teeth (1.6, 2.1, 2.4, 3.6, 4.1 and 4.4). Data were obtained from the neighbouring tooth in cases where one of these teeth were not present. Deciduous teeth and teeth with developmental disturbances were excluded. Regarding ETW, prevalence and severity was recorded using the Basic Erosive Wear Examination (BEWE index). According to this index, every permanent tooth surface is evaluated and is classified into a 4 score criteria, "0" being an indication for the absence of ETW, "1" being initial loss of surface texture, "2"* being distinct defect, hard tissue loss affecting less than 50% of tooth surface and "3"* being an indication for hard tissue loss and presence of ETW in more than the 50% of the surface (*usually involving dentin). The final BEWE sum score was the result of the sum of the highest score recorded per sextant .

Reproducibility Two paediatric dentists (FM and SD) were educated, instructed and calibrated for DMFT index. The examiners scored twice several clinical cases in two sessions separated by a two-week period. Then, the examiners scores were compared against an experienced benchmark (LM).

Questionnaire A validated questionnaire was applied in order to assess oral hygiene and dietary habits. Prior to initiation of the study, a content validation of the questionnaire was performed by five professors with experience in epidemiology. For the reliability of the questionnaire, a group of 20 students (15-year-old) were asked to complete the questionnaire twice separated by a two-week period. Once validated, the questionnaire was applied to each participant of the study on the same day of dental examination. Participants were asked to answer the questionnaire according to their habits just before they enter the rehabilitation centre.

ELIGIBILITY:
Inclusion Criteria:

* obesity in case group (having a BMI above the 97th percentile + 2.17 to+2.18 SDS),
* normal weight in the control group (BMI between the 10th and 90th percentile -1.64 to +1.64 SDS). Obese and normal weight groups were defined using the BMI according to the European Childhood Obesity Group (ECOG) and the growth curves for Flemish boys and girls (2-20years).

Exclusion Criteria:

* smoking
* chronic disease
* receive treatment with antibiotics three months prior to the study
* consume medications with side effects on the gums
* wearing orthodontic appliances
* other ethnicity (not Belgian) were excluded as ethnicity is an influential factor in the relation between caries and obesity.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cases were all the obese children/adolescents (N=81; age range 11 to 18 years-old) who were recently participating in a treatment program for obese patients in a rehabilitation centre for chronic diseases (Zee Preventorium, De Haan, Belgium). Based on the number of cases, 81 normal weight students of two Belgian secondary schools (Deinze, Belgium) were recruited as controls. Controls were sex-age-matched, had the same education level and socioeconomic status (SES).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-10-25 (Actual); Study Completion 2015-10-25 (Actual)

PRIMARY OUTCOMES:
Oral health status | Once on the day of dental examination
  Caries experience was screened using DMFT index (Decayed, Missing, Filled Teeth) with a subdivision for D1 (early caries, 'white spots'), D2 (enamel caries) or D3 (dentine caries). The periodontal status was evaluated by measuring the Gingivitis index (Silness and Loë, 1963), Plaque index (Silness and Loë, 1964) and the presence of periodontal pockets (≥4mm) in all Ramfjord teeth (1.6, 2.1, 2.4, 3.6, 4.1 and 4.4). Data were obtained from the neighbouring tooth in cases where one of these teeth were not present. Deciduous teeth and teeth with developmental disturbances were excluded. Regarding ETW, prevalence and severity was recorded using the Basic Erosive Wear Examination (BEWE index).
Association of oral health status and diet/oral hygiene habits | Once on the same day of dental examination
  A validated questionnaire was applied in order to assess oral hygiene and dietary habits. The questionnaire was applied to each participant of the study on the same day of dental examination. Participants were asked to answer the questionnaire according to their habits just before they enter the rehabilitation centre.

IPD SHARING:
Plan to Share IPD: No